CLINICAL TRIAL: NCT04228822
Title: Safety and Feasibility of a Low Carbohydrate Diet in Children With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: ICTS BJH (Unknown); Center for Diabetes Translation Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201911121
Record Dates: First submitted 2019-12-11; First posted 2020-01-14 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Intervention Model Description: 20 participants will be randomized to the intervention group (low carbohydrate diet) and 20 participants will be randomized to the control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low carb diet intervention group (Experimental): Low carbohydrate diet defined as 25-35% of total energy intake
  Interventions: Other: Low carbohydrate diet
- Control (No Intervention): Standard diet defined as 45-65% total energy intake

INTERVENTIONS:
Other: Low carbohydrate diet — 25-35% of carbohydrates from total energy intake
  Arms: Low carb diet intervention group

SUMMARY:
Good glycemic control in individuals with Type 1 diabetes (T1D), has been proven to reduce the risk of diabetes-related complications. Despite technological advances such as the use of insulin delivery devices and continuous glucose monitoring, the average glycemic control in T1D is poor. Though dietary management plays a major role in the overall management of T1D, and it is often classified as the most challenging aspect of treatment, the 2019 Standards of Medical Care in Diabetes for children and adolescents do not clearly address dietary management. As carbohydrate is the macronutrient with the greatest impact on blood glucose, it is reasonable to suggest that carbohydrate reduction will minimize postprandial glucose excursions and improve diabetes control. For this reason, low carbohydrate diets (LCD) have gained popularity, and observational studies report positive glycemic outcomes. However, to date, scientific evidence from randomized trials on the impact of LCD in children with T1D is lacking. Thus, the over-arching goal of this pilot study is to evaluate the feasibility and safety of a low carbohydrate diet in children with T1D, and as an exploratory aim, we will evaluate the efficacy of LCD on glycemic control.

DETAILED DESCRIPTION:
The investigators aim to study 40 subjects ages 5-11 with T1D to evaluate the feasibility of LCD. Participants will be asked to attend a total of 5 visits (4 in person and 1 phone visit) during the 6 month-duration of the study. Participants will be randomized to an intervention group with a LCD (50% of carbohydrate recommended daily allowance) vs. the standard diet.

During the screening visit, participants will be assessed by a dietitian to categorize their existing dietary regimen before randomization to either the LCD or the standard diet. In addition, participant's insulin regimen (either pump settings or multiple dose insulin injection therapy) will be reviewed for insulin dose adjustments as needed over a 2 week-period.

ELIGIBILITY:
Inclusion Criteria:

* Patients 5-11 years of age, with history of Type 1 diabetes for longer than 2 years,
* No carbohydrate restrictions at the time of recruitment.
* No medications that could affect appetite
* Regular attendance at the clinic (3-4 times per year),
* Glycated hemoglobin (HbA1c) <10%.

Exclusion Criteria:

* Impaired renal or liver function,
* Chronic seizures or global developmental delay,
* Diagnosed with ADHD and/or on ADHD medications
* Use of drugs other than insulin affecting glucose metabolism
* Severe eczema
* Celiac disease

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Number of hypoglycemic events | 6 month study period
  Using a continuous glucose monitor (CGM) and home glucose meter, investigators will calculate the number of hypoglycemic events (glucose values <70 mg/dL but ≥ 54 mg/dL and those <54 mg/dL), number of severe hypoglycemia and time spent in hypoglycemia (values <70 mg/dL but ≥ 54 mg/dL and <54 mg/dL).
Episodes of diabetes related visits to the hospital, DKA | 6 month study period
  Investigators will obtain data prospectively from medical records and will estimate the frequency of DKA, diabetes related hospitalizations / emergency department visits.
Dyslipidemia | 6 month study period
  Investigators will evaluate the changes in LDL levels among the study groups.

SECONDARY OUTCOMES:
Glycemic control | 6 month duration of the study
  Investigators will evaluate the changes in glycemic control among the groups using HbA1c at baseline, 3 and 6 months.
Glucose variability | 6 month study period
  Using CGM data investigators will evaluate glucose variability using standard deviation (SD) of all glucose values. Secondary endpoints will include time of the day spent in range (values between 70-140 mg/dl and between 70 and 180mg/dl), in hypoglycemia (values <70 mgl/dl but ≥ 54 mg/dl and <54 mg/dl) and in hyperglycemia (values >180mg/dl and >250 mg/dl).

CONTACTS AND LOCATIONS:
Locations (1):
- St Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No